CLINICAL TRIAL: NCT04943835
Title: Validity of a Test of Functional Cognition in Persons With Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1607017448
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational - No intervention

SUMMARY:
The purpose of this study is to test the validity of the Weekly Calendar Planning Activity (WCPA), a test of functional cognition in persons with acquired brain injury. We will formally examine the utility, baseline profile and validity of the WCPA with adults ages 21 and above with acquired brain injury for both the WCPA 17 and WCPA 10 versions.

DETAILED DESCRIPTION:
The purpose of this study is to test the validity of the Weekly Calendar Planning Activity (WCPA), a test of functional cognition in persons with acquired brain injury. We will formally examine the utility, baseline profile and validity of the WCPA with adults ages 21 and above with acquired brain injury for both the WCPA 17 and WCPA 10 versions. The Weekly Calendar Planning Activity (WCPA) is a performance-based Cognitive Instrumental activities of daily living (C-IADL) task that requires working memory, planning, shifting, inhibition, and self-monitoring. The WCPA requires the examinee to input a series of 10 appointments, into a mock weekly calendar/schedule while following multiple rules, managing appointment conflicts, ignoring distracting questions by the examiner and keeping track of time. The WCPA is used routinely by occupational therapists for those with acquired brain injury, during their stay on the inpatient rehabilitation unit, prior to discharge as a measure of IADL. Persons who are currently receiving occupational therapy and would typically be given the WCPA within the course of routine occupational therapy, will be asked for permission to include their results within a database for the project. Persons who are alert, oriented x3, able to attend for at least 10 minutes, are able to read and write legibly in English would typically be administered the WCPA. Potential participants will be identified by their primary therapist. If the person does not provide consent, the WCPA will be administered as part of usual care but the results will not be included within the project.

ELIGIBILITY:
Inclusion Criteria:

* Able to attend for at least 10 minutes
* Able to read and write legibly in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with acquired brain injury receiving inpatient occupational therapy
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
WCPA Percent Accuracy | During hospitalization, approximately one week
  The Weekly Calendar Planning Activity (WCPA) is a performance-based Cognitive Instrumental activities of daily living (C-IADL) task that requires working memory, planning, shifting, inhibition, and self-monitoring. The WCPA requires the examinee to input a series of 10 appointments, into a mock weekly calendar/schedule while following multiple rules, managing appointment conflicts, ignoring distracting questions by the examiner and keeping track of time. WCPA percent accuracy is the number of appointments entered correctly out of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Dell, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No